CLINICAL TRIAL: NCT00993694
Title: Dapsone Induced Methemoglobinemia in Pediatric Hematologic Malignancy and Aplastic Anemia
Brief Title: Methemoglobinemia in Young Patients With Hematologic Cancer or Aplastic Anemia Treated With Dapsone
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Esbenshade, Assistant Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: CDR0000652603; P30CA068485 (NIH); VU-VICC-PED-0916; IRB# 090009; NCT00960050 (obsolete NCT alias)
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorder; Methemoglobinemia; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Nonmalignant Neoplasm
Keywords: methemoglobinemia; aplastic anemia; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; juvenile myelomonocytic leukemia; mast cell leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related lymphoblastic lymphoma; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; recurrent/refractory childhood Hodgkin lymphoma; stage I childhood Hodgkin lymphoma; stage II childhood Hodgkin lymphoma; stage IV childhood Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage II childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; Burkitt lymphoma; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; childhood nasal type extranodal NK/T-cell lymphoma; intraocular lymphoma; primary central nervous system non-Hodgkin lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; essential thrombocythemia; polycythemia vera; extramedullary plasmacytoma; isolated plasmacytoma of bone; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; primary systemic amyloidosis; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; childhood myelodysplastic syndromes; recurrent childhood anaplastic large cell lymphoma; stage I childhood anaplastic large cell lymphoma; stage II childhood anaplastic large cell lymphoma; stage III childhood anaplastic large cell lymphoma; stage IV childhood anaplastic large cell lymphoma; stage III childhood Hodgkin lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Lymphoproliferative Disorders; Methemoglobinemia; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Neoplasms; Anemia, Aplastic; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Recurrence; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Extranodal NK-T-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis | interventions — Drug Therapy; Dapsone

INTERVENTIONS:
Drug: chemotherapy
Drug: dapsone
Other: medical chart review
Procedure: assessment of therapy complications

SUMMARY:
RATIONALE: Gathering information about how often methemoglobinemia occurs in young patients receiving dapsone for hematologic cancer or aplastic anemia may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This research study is looking at methemoglobinemia in young patients with hematologic cancer or aplastic anemia treated with dapsone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the incidence of methemoglobinemia in patients with hematologic malignancy or aplastic anemia who received dapsone prophylaxis through a retrospective chart review encompassing the last 15 years.
* Identify major risk factors for developing methemoglobinemia.

OUTLINE: Medical charts are reviewed. Of particular interest is demographic information, reasons for beginning dapsone prophylaxis, duration of dapsone prophylaxis, dapsone dosing, methemoglobin level, and treatment with methylene blue.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematologic malignancy or aplastic anemia

  * Treated within the past 15 years with dapsone prophylaxis during treatment of primary disease

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of methemoglobinemia in patients with hematologic malignancy or aplastic anemia who received dapsone prophylaxis through a retrospective chart review encompassing the last 15 years
Major risk factors for developing methemoglobinemia

CONTACTS AND LOCATIONS:
Overall Officials: Adam J. Esbenshade, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee